CLINICAL TRIAL: NCT00594360
Title: Exercise on Prescription: Effects and Comparison of Psychological Parameters Physical Activity, Physical Fitness, and Health Physical Between Participants in a Danish Version of Exercise on Prescription.
Brief Title: Evaluation of Effect of Exercise on Prescription - a Psychological Perspective
Acronym: EoP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: The County of Funen, Denmark (Other Government); The County of Frederiksberg (Unknown); National Board of Health, Denmark (Other Government)
Responsible Party: Gitte Halling, Faculty of Health Sciences, University of Southern Denmark, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36/154-150775; 2005-41-5248
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2007-12

CONDITIONS: Physical Inactivity; Motivation; Behavior Change
Keywords: Exercise Prescription; Self-efficacy; Decisional Balance; Readiness to Change; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Behavioral: Exercise on Prescription

INTERVENTIONS:
Behavioral: Exercise on Prescription — Exercise two times a week for two months at a physiotherapist. Afterwards exercise one time a week at a physiotherapist and self-contained training one time a week for 2 months.
  Other Names: Open Label, Active Control, Efficacy Study, Best practice

SUMMARY:
The purpose of this study is to evaluate the effect of a primary healthcare intervention called 'Exercise on Prescription' aimed at increasing level of physical activity and psychological parameters in a population of sedentary patients with increased risk of developing lifestyle diseases. The effect is evaluated using patient-reported variables.

DETAILED DESCRIPTION:
Exercise prescriptions are used for initiating a physical active lifestyle in sedentary populations.

A Danish project called 'Exercise on Prescription' (EoP) is implemented in primary healthcare. Patients eligible for EoP are non-institutionalised adults with medically controlled lifestyle diseases or risk factors of lifestyle diseases, who are motivated to change lifestyle, able to improve health status through a physical active lifestyle, and willing to pay a fee of €100 for the intervention.

The purpose of this study is to assess the effect on: 1) Self-efficacy, 2) Readiness to change, 3) Decisional balance, 4) physical activity level, and 5) health related quality of life.

The EoP-group is compared to an intervention group receiving only motivational counselling.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the Exercise on Prescription scheme by their general practitioner
* Volunteer to participate in the trial

Exclusion Criteria:

* BMI over 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-11; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Self-efficacy level at 4, 10 and 16 months. Patient-reported Decisional balance level at 4, 10 and 16 months. Patient-reported Readiness to change level at 4, 10 and 16 months. | 16 months

SECONDARY OUTCOMES:
Patient-reported physical activity level at 4, 10 and 16 months. . Patient-reported health related quality of life at 4, 10 and 16 months. Patient-reported compliance with national guidelines for physical activity at 4, 10 and 16 months. | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Lis Puggaard, PhD, Principal Investigator — Centre of Applied and Clinical Exercise Science, Institute of Sport Sciences and Clinical Biomechanics, University of Southern Denmark, Denmark
Locations (1):
- Centre of Applied and Clinical Exercise Science, Institute og Sport Sciences and Clinical Biomechanics, University of Southern Denamrk, Odense, Denmark

REFERENCES:
- [Derived] Bredahl TV, Puggaard L, Roessler KK. Exercise on Prescription. Effect of attendance on participants' psychological factors in a Danish version of Exercise on Prescription: a study protocol. BMC Health Serv Res. 2008 Jun 26;8:139. doi: 10.1186/1472-6963-8-139. PMID 18582371